CLINICAL TRIAL: NCT01672697
Title: Effects of Physical Therapy on Pelvic Floor Symptoms and Quality of Life in Postpartum Women Following Severe Perineal Trauma: a Randomized Controlled Trial
Brief Title: Physical Therapy for Women With Obstetric Trauma and Anal Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 12005-TriHealth
Record Dates: First submitted 2012-08-21; First posted 2012-08-27 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2017-03

CONDITIONS: Sphincter Ani Incontinence; Obstetric Trauma
Keywords: anal incontinence; genital trauma; physical therapy; anal manometry
MeSH Terms: conditions — Encopresis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical & Behavioral Therapy Group (Experimental): Intervention Group: Randomized to Physical Therapy (PT)
  1. 2-week visit which includes: Demographic Data, Physical Exam, ehavioral Therapy (BT) handouts Functional questionnaires administered Physiologic measurements obtained
  2. Follow-up Evaluation-6-week visit PT session #1 Functional questionnaires administered
  3. Follow-up Evaluation-8-week visit PT session #2
  4. Follow-up Evaluation-10-week visit PT session #3
  5. Study Completion Visit-12-week visit Functional questionnaires administered PT session #4 Physiologic measurements Physical Exam
  6. Long-term Follow-up-24-weeks Functional questionnaires administered by mail
  Interventions: Behavioral: Physical Therapy (PT) and Behavioral Therapy (BT)
- Control Group (No Intervention): Control Group:
  1. Baseline Data obtained at 2-week visit Demographic Data General Physical Exam findings Functional questionnaires administered in person (FIQOL, FISI, SF-12, FSFI, UDI-6, IIQ-7) Physiologic measurements obtained (Vaginal EMG, Anal-rectal manometry)
  2. Follow-up Evaluation at 6-week visit Functional questionnaires administered in person at patient's previously scheduled postpartum office visit with primary Ob/Gyn or by mail
  3. Study Completion Visit at 12-week visit Functional questionnaires administered Physiologic measurements obtained Physical Exam findings
  4. Long-term Follow-up at 24-weeks - Functional questionnaires administered by mail

INTERVENTIONS:
Behavioral: Physical Therapy (PT) and Behavioral Therapy (BT) — 1. Physical Therapy (PT) Protocol states that each participant in the treatment arm only will undergo a total of four 45-minute sessions with a certified pelvic floor (PF) physical therapist over the course of the 12 weeks. Routine monitoring of patient progress will be performed. Each session includes using the body core muscles and internal pelvic floor muscles, focusing on PF protection techniques, PF exercises, Core exercises, progression to full ADLs(activities of daily living), and an exercise routine.
  2. Behavioral Therapy (BT) Instructions are given only to participants in the treatment arm after randomization at week-2 visit; handout provides specific instructions about appropriate diet, hygiene and level of activity during the 12 weeks of enrollment.
  Other Names: Internal Pelvic Floor Physical Therapy
  Arms: Physical & Behavioral Therapy Group

SUMMARY:
Our primary objective is to determine if physical therapy (PT) and behavioral therapy (BT) in the post-partum period after a vaginal delivery complicated by genital trauma help to improve a woman's quality of life, specifically in regard to anal incontinence. To be able to study this, the investigators need to know how well the muscles of a woman's pelvic floor function after a vaginal delivery and this requires measuring their strength during a pelvic exam. At present, there are no studies that have looked at whether the intervention of PT/BT improves a woman's anal incontinence quality of life after sustaining genital trauma during vaginal deliveries

DETAILED DESCRIPTION:
This is a prospective trial involving 65 woman who sustained a severe laceration or episiotomy during their first vaginal delivery to determine if postpartum intervention with physical/behavioral therapy improves their quality of life in regard to anal incontinence. The primary outcome measure is functional and based on a change in score of the Fecal Incontinence Quality of Life (FIQOL) validated questionnaire from baseline (2-weeks after delivery date) to study completion (12-weeks after delivery date). The secondary outcome measure is physiologic and reflects a change in anal sphincter resting tone from baseline to study completion.

After the screening questionnaires to determine eligibility in the study, each study subject will be consented for participation then undergo a baseline physical exam (including pelvic exam and rectal exam) at a range of 2- to 4- weeks after delivery date. In addition, after this initial exam, all women will be randomized immediately to receive (1) no further treatments, or (2) physical and behavioral therapy.

The investigators will study these two groups of women for 24 total weeks after the date of delivery. The intervention group will include patients randomized to receiving PT/BT for 4 weekly sessions after their vaginal delivery and laceration (episiotomy) repair. The control group (no intervention) will include patients randomized to receiving the standard of care (no physical or behavioral therapy) after their vaginal delivery and laceration (episiotomy) repair.

Each group will undergo the baseline testing: a pelvic exam (to measure the strength of your muscles) and anal-rectal manometry (i.e. rectal exam with insertion of a small sensor to measure the strength of your sphincter); and be asked to complete a series of brief questionnaires. These questionnaires will be administered again to both groups at 6-weeks, 12-weeks, and 24-weeks after their delivery date. Study completion physical exams including a repeat pelvic exam and repeat anal-rectal manometry will be conducted at 12-weeks after delivery date.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women aged 18 years of older
* Vaginal delivery, vacuum-assisted-vaginal-delivery (VAVD), or forceps-assisted-vaginal-delivery (FAVD) of a neonate of gestational age:
* 27 completed weeks
* Singleton or vaginal delivery of multiple gestation
* Able to read and speak the English language

Exclusion Criteria:

* Unable to comply with physical therapy or office visits
* Unreliable transportation
* Preexisting neurologic, musculoskeletal or neuromuscular disorder rendering them unable to perform physical therapy requirements
* Cesarean delivery
* History of prior surgery for anorectal incontinence (i.e. sphincteroplasty

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-09-12 (Actual); Primary Completion 2016-03-17 (Actual); Study Completion 2016-03-17 (Actual)

PRIMARY OUTCOMES:
Fecal Incontinence Quality of Life (FIQOL) | baseline (2-weeks post delivery) to completion (12-weeks post delivery)
  The Fecal Incontinence Quality of Life Scale (FIQOL) is a 29-item instrument developed with the support of the American Society of Colon and Rectal Surgeons that measures the impact of anal incontinence over four domains: Lifestyle, Coping/behavior, Depression/self-perceptions, and Embarrassment. The FIQL has demonstrated validity and reliability.

SECONDARY OUTCOMES:
Anal-rectal manometry (ARM) | baseline (2 weeks post delivery) to completion (12 weeks post delivery)
  Anal Rectal Manometry (ARM) will be completed by all participants at baseline (week 2 visit) and completion (week 12 visit); a small caliber soft flexible disposable air-filled catheter will be placed in the patient's rectum to a depth of 5cm in order to obtain the resting tone and squeezing pressure of the sphincter, per the protocol and patient preparatory instructions as provided by Laborie Medical Technologies (Mississauga, Ontario, Canada) for use with their Triton Aquarius Urodynamics® chair and compatible UDS120 software.

OTHER OUTCOMES:
Fecal Incontinence Severity Index (FISI) | baseline (2-weeks post delivery) to completion (12-weeks post delivery)
  The Fecal Incontinence Severity Index (FISI) is a frequency matrix developed with support of the American Society of Colon and Rectal Surgeons that assigns patient-weighted values to various frequencies and types of incontinence. The FISI has demonstrated correlation with the FIQL.
Short Form-12 (SF-12) | baseline (2-weeks post delivery) to completion (12-weeks post delivery)
  The Short Form-12 (SF-12) is a brief 12-item questionnaire to assess a subject's current general health.
Female Sexual Function Index (FSFI) | baseline (2-weeks post delivery) to completion (12-weeks post delivery)
  The Female Sexual Function Index (FSFI) is a 19-item questionnaire that can be administered in any age group and focuses on individual function via six domains: desire, arousal, lubrication, orgasm, satisfaction and pain.
Urogenital Distress Inventory (UDI-6) | baseline (2-weeks post delivery) to completion (12-weeks post delivery)
  The Urogenital Distress Inventory-6 (UDI-6) is a 6-question instrument about lower urinary tract symptoms separated into 3 scales: irritative symptoms, obstructive/discomfort symptoms and stress symptoms. Respondents rate the degree to which each is bothersome on a 4-point scale.
Incontinence Impact Questionnaire-7 (IIQ-7) | baseline (2-weeks post delivery) to completion (12-weeks post delivery)
  The Incontinence Impact Questionnaire-7 (IIQ-7) is a 7 item companion to the UDI-6 with condition-specific quality of life questions assessing the degree to which lower urinary tract symptoms affect daily activities via 4 scales: travel, social, emotional and physical.
Vaginal Electromyography (EMG) | baseline (2-weeks post delivery) to completion (12-weeks post delivery)
  Vaginal EMG readings will be completed by all participants at baseline (week 2 visit) and completion (week 12 visit); these electrodes are inserted vaginally and readings are recorded in μV to determine pelvic floor tone for correlation with ARM in order to determine if differences in primary and secondary outcomes for both groups are due to the BT/PT intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pauls, MD, Study Director — TriHealth Inc.
Locations (1):
- TriHealth, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Woodley SJ, Lawrenson P, Boyle R, Cody JD, Morkved S, Kernohan A, Hay-Smith EJC. Pelvic floor muscle training for preventing and treating urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2020 May 6;5(5):CD007471. doi: 10.1002/14651858.CD007471.pub4. PMID 32378735
- [Derived] Oakley SH, Ghodsi VC, Crisp CC, Estanol MV, Westermann LB, Novicki KM, Kleeman SD, Pauls RN. Impact of Pelvic Floor Physical Therapy on Quality of Life and Function After Obstetric Anal Sphincter Injury: A Randomized Controlled Trial. Female Pelvic Med Reconstr Surg. 2016 Jul-Aug;22(4):205-13. doi: 10.1097/SPV.0000000000000255. PMID 26829343